CLINICAL TRIAL: NCT06166836
Title: A Phase 1b/II, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of D-1553 Combined With IN10018 in Subjects With Locally Advanced or Metastatic Solid Tumors With KRAS G12C Mutation
Brief Title: a Study to Evaluate the Safety and Efficacy of D-1553 Combined With IN10018 in KRAS G12C Mutant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Collaborators: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1553-106/IN10018-602
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1b-Dose Escalation Part (Experimental): To evaluate the safety and Recommended Phase 2 dose (RP2D) of D-1553 in combination with IN10018 in previously-treated solid tumors.
  Interventions: Drug: D1553; Drug: IN10018（Ifebemtinib）
- Phase II Cohort A-previously-treated CRC with KRAS G12C mutation（Treatmnt Group） (Experimental): To evaluate the safety and antitumor efficacy of D-1553 in combination with IN10018 in previously-treated CRCs with KRAS G12C mutation.
  Interventions: Drug: D1553; Drug: IN10018（Ifebemtinib）
- Phase II Cohort A-previously-treated CRC with KRAS G12C mutation (Control Group) (Active Comparator): To evaluate the safety and antitumor efficacy of D-1553 in previously-treated CRCs with KRAS G12C mutation.
  Interventions: Drug: D1553
- Phase II Cohort B-treatment-naïve or previously-treated NSCLC with KRAS G12C mutation (Experimental): To evaluate the safety and antitumor efficacy of D-1553 in combination with IN10018 in advanced NSCLCs with KRAS G12C mutation.
  Interventions: Drug: D1553; Drug: IN10018（Ifebemtinib）
- Phase II Cohort C-other previously-treated solid tumors with KRAS G12C mutation (Experimental): To evaluate the safety and antitumor efficacy of D-1553 in combination with IN10018 in other solid tumors with KRAS G12C mutation
  Interventions: Drug: D1553; Drug: IN10018（Ifebemtinib）

INTERVENTIONS:
Drug: D1553 — D1553 orally taken，600mg twice a day
Drug: IN10018（Ifebemtinib） — IN10018 orally taken once daily at approximately the same time each day
  Other Names: BI 853520
  Arms: Phase 1b-Dose Escalation Part; Phase II Cohort A-previously-treated CRC with KRAS G12C mutation（Treatmnt Group）; Phase II Cohort B-treatment-naïve or previously-treated NSCLC with KRAS G12C mutation; Phase II Cohort C-other previously-treated solid tumors with KRAS G12C mutation

SUMMARY:
This is a phase 1b/II, open-label study to evaluate the safety, tolerability, pharmacokinetics and antitumor activities of D-1553 in combination with IN10018 in subjects with locally advanced or metastatic solid tumor with KRAS G12C mutation.

DETAILED DESCRIPTION:
This study includes 2 phases: Phase Ib-Dose Escalation and Phase II-Dose Expansion. Phase Ib-Dose Escalation part will enroll at least 6 subjects to identify the safety and RP2D of D1553 in combination with IN10018 in KRAS G12C mutant solid tumors. Phase II-Dose Expansion part contains 3 cohorts with cohort A to enroll advanced colorectal cancer (CRC) with KRAS G12C mutation, cohort B to enroll advanced non-small cell lung cancer (NSCLC) with KRAS G12C mutation, and cohort C to enroll other advanced solid tumors with KRAS G12C mutation. Phase II study is to evaluate the safety and antitumor activities of D-1553 in combination with IN10018 in KRAS G12C mutant solid tumors. The sample size in each cohort is estimated per Simon's 2-stage design. In Cohort A, when Simon's 2-stage study achieved statistical hypothesis, an open-label, randomized study will be conducted for factorial analysis to evaluate the contribution of IN10018 in the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥ 18 years at the time of signing the informed consent form.
2. Subjects with pathologically confirmed locally advanced or metastatic solid tumors.
3. Confirmed positive KRAS G12C mutation in tumor tissue or other biospecimens (only for phase1b) containing cancer cells or DNA.
4. Tumor types in different phases and cohorts: 1) Phase 1b: subjects with locally advanced or metastatic solid tumors who have progressed on or failed in standard therapy, and no standard treatment is available. 2) Phase II Cohort A: subjects with locally advanced or metastatic CRC. 3) Phase II Cohort B: subjects with locally advanced or metastatic NSCLC. 4) Phase 2 Cohort C: subjects with other locally advanced or metastatic solid tumors.
5. Has measurable lesions at baseline according to RECIST 1.1 criteria.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate bone marrow, liver, renal, and coagulation function within 7 days prior to the first dose.

Exclusion Criteria:

1. Prior KRAS G12C inhibitors treatment.
2. Have known symptoms of spinal cord compression, instable or symptomatic central nervous system (CNS) metastases, and/or carcinomatous meningitis.
3. Have a history of stroke or other serious cerebrovascular diseases within 12 months prior to the first dose.
4. Have had interstitial lung disease or any active infection requiring systemic treatment within 14 days prior to the first dose.
5. Has a history of severe cardiovascular disease such as acute myocardial infarction, severe/unstable angina, QTc prolongation, or poorly controlled hypertension.
6. Haven't recovered from toxicity due to prior antitumor therapy
7. Pregnant or lactating women.
8. Malignant neoplasms other than study disease within 5 years prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of D1553 in combination with IN10018 in solid tumors with KRAS G12C mutation | Through study completion, approximately 3 years
  Evaluate the number of patients with dose-limited toxicities (DLTs); Determine the RP2D of D1553 in combination with IN10018 in solid tumors with KRAS G12C mutation.
Objective Response Rate (ORR) of D1553 in combination with IN10018 in solid tumors with KRAS G12C mutation | Through study completion, approximately 3 years
  Defined as the proportion of subjects with complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-free Survival (PFS) of D1553 in combination with IN10018 in solid tumors with KRAS G12C mutation | Through study completion, approximately 3 years
  Defined as the time from the first dose of study treatment to first documentation of disease progression or to death due to any cause, whichever comes first.
Duration of Response (DoR) of D1553 in combination with IN10018 in solid tumors with KRAS G12C mutation | Through study completion, approximately 3 years
  Defined as the time from start of the first documentation of CR or PR to the first documentation of disease progression or to death due to any cause, whichever comes first.
Disease Control Rate (DCR) of D1553 in combination with IN10018 in solid tumors with KRAS G12C mutation | Through study completion, approximately 3 years
  Defined as the proportion of patients with CR, PR, or stable disease (SD).
Overall survival (OS) of D1553 in combination with IN10018 in solid tumors with KRAS G12C mutation | Through study completion, approximately 3 years
  Defined as the time from the first dose of study treatment to the date of death due to any cause.
Number of subjects with adverse event | Through study completion, approximately 3 years
  The number of subjects who experienced AEs is presented.
Plasma concentrations of D-1553 and IN10018 in solid tumors with KRAS G12C mutation | Through study completion, approximately 3 years
  Plasma concentrations of D-1553 and IN10018
PK: Cmax of D-1553 and IN10018 | Through study completion, approximately 3 years
  Maximum concentration (Cmax)
PK: Cmin of D-1553 and IN10018 | Through study completion, approximately 3 years
  Minimum concentration (Cmin)
PK:t1/2 of D-1553 and IN10018 | Through study completion, approximately 3 years
  Elimination half-life (t1/2).
PK:CL/F of D-1553 and IN10018 | Through study completion, approximately 3 years
  apparent clearance (CL/F)
PK:Vd/F of D-1553 and IN10018 | Through study completion, approximately 3 years
  Apparent volume of distribution (Vd/F)
PK: AUC of D-1553 and IN10018 | Through study completion, approximately 3 years
  Area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Zhengbo Song, Principal Investigator — Study Principal Investigator
Locations (10):
- China (10):
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Hunan Cancer Hospital, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - General Hospital Of Eastern Theater Command, Nanjing
  - Renmin Hospital of Wuhan University, Wuhan
  - Xuzhou Central Hospital, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The first Affiliated Hospital of Zhengzhou University, Zhengzhou